CLINICAL TRIAL: NCT03066739
Title: Effect of Ultra-low Dose Naloxone on Remifentanil-Induced Hyperalgesia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated early due to low enrollment. Only 8 participants enrolled out of the target 105.
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Ariana M. Nelson, Associate Clinical Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20141345
Record Dates: First submitted 2017-02-21; First posted 2017-02-28 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Hyperalgesia
MeSH Terms: conditions — Hyperalgesia | interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- LO-low dose remifentanil (Active Comparator): low dose remifentanil (LO, 0.1 micrograms/kg/mL),
  Interventions: Drug: Remifentanil
- HI-high dose remifentanil with placebo (Active Comparator): high dose remifentanil (0.4 mg) combined with placebo (HI, 0.4 micrograms/kg/mL)
  Interventions: Drug: Remifentanil+ Placebo
- HN-high dose remifentanil with ultra-low dose naloxone (Active Comparator): high dose remifentanil (0.4 mg) combined with ultra-low dose naloxone (HN, 0.004 micrograms/kg/mL naloxone).
  Interventions: Drug: Remifentanil +ultra-low dose naloxone

INTERVENTIONS:
Drug: Remifentanil — 0.1 micrograms/kg/mL
  Other Names: LO
  Arms: LO-low dose remifentanil
Drug: Remifentanil+ Placebo — high dose remifentanil (0.4 mg) combined with placebo (HI, 0.4 micrograms/kg/mL)
  Other Names: HI
  Arms: HI-high dose remifentanil with placebo
Drug: Remifentanil +ultra-low dose naloxone — high dose remifentanil (0.4 mg) combined with ultra-low dose naloxone (HN, 0.004 micrograms/kg/mL naloxone
  Other Names: HN
  Arms: HN-high dose remifentanil with ultra-low dose naloxone

SUMMARY:
The purpose of this study is to evaluate whether using ultra-low dose naloxone, an opioid antagonist, has the potential to block remifentanil-induced hyperalgesia and tolerance following surgery.

There are 3 study groups: (1) low dose remifentanil (LO, 0.1 micrograms/kg/mL), (2) high dose remifentanil (0.4 mg) combined with placebo (HI, 0.4 micrograms/kg/mL), or (3) high dose remifentanil (0.4 mg) combined with ultra-low dose naloxone (HN, 0.004 micrograms/kg/mL naloxone).

The hypothesis of the study is that occurrence of remifentanil-induced hyperalgesia (low score in mechanical pain threshold) in the HN group will be lower than in the HI group.

DETAILED DESCRIPTION:
Purpose:

Opioid antagonists at ultra-low doses have been used with opioid agonists to prevent or limit opioid tolerance. Remifentanil, a rapid onset/offset opioid that is often used as an anesthesia adjunct intraoperatively, has been associated with the development of hyperalgesia and opioid tolerance postoperatively. Opioid-induced hyperalgesia (OIH) induced by remifentanil intraoperatively may be a factor contributing to an increase in postoperative pain as well as difficulty in controlling such pain. The purpose of this study will be to evaluate whether an ultra-low dose of naloxone, an opioid antagonist, could block remifentanil-induced hyperalgesia and tolerance following surgery.

This research will help elucidate the degree of OIH after surgeries involving remifentanil and determine if a new technique can be employed to decrease remifentanil-induced OIH. By mitigating OIH, patients should have a decrease in postoperative pain and an increase in patient satisfaction at UCI and other hospitals where such a technique is employed.

There are 3 study groups: (1) low dose remifentanil (LO, 0.1 micrograms/kg/mL), (2) high dose remifentanil (0.4 mg) combined with placebo (HI, 0.4 micrograms/kg/mL), or (3) high dose remifentanil (0.4 mg) combined with ultra-low dose naloxone (HN, 0.004 micrograms/kg/mL naloxone).

Background:

Opioid-induced hyperalgesia is a paradoxical increase in pain sensitivity following opioid exposure. The mechanism for this is likely due to an alteration in opioid receptor signaling with disruption of G-protein coupling and opioid-induced activation and hypertrophy of spinal glial cells (gliosis). Opioid-induced hyperalgesia has been noted with many different opioids, and the most well documented hyperalgesic effect is with remifentanil.

Various agents have been used in an attempt to reduce the development hyperalgesia following remifentanil. While there are few reports on the effect of ultra-low dose naloxone on opioid-induced hyperalgesia, recent evidence is emerging regarding its use in pain management. Ultra-low dose naloxone has been shown to prevent remifentanil-induced pain hypersensitivities (allodynia and hyperalgesia) in rats. However, there are little to no studies on reducing the adverse effects of remifentanil with naloxone in human subjects.

Existing knowledge and previous research:

Attempts have been made with various agents to reduce the development of tolerance and hyperalgesia following remifentanil. Postoperative hyperalgesia and its prevention has been studied with ketamine , Magnesium , Gabapentin, Clonidine, Lornoxicam , Dextromethorphan , Paracetamol , Morphine , Dexmedetomidine , Adenosine, COX inhibitors , Amantadine , Nitrous oxide, Fentanyl, Pregabalin , Buprenorphine, Midazolam, Dexamethasone. Relevant to our current hypothesis is the report that concomitant administration of ultra-low dose naloxone and naltrexone with remifentanil prevented OIH. However, there are no studies on reducing the adverse effects of remifentanil with ultra-low dose naloxone in human subjects.

While the traditional role of opiate antagonists have been in cases of opioid overmedication, recent evidence is emerging regarding their use in pain management. Gan et al. 1997 used an ultra-low dose naloxone infusion (0.00025 mg/kg/h or 0.001 mg/kg/h) in postoperative patients receiving IV morphine via a patient-controlled analgesia (PCA) device. Good pain relief was experienced in all groups, however consumption of PCA morphine was significantly reduced in patients that received the lowest infusion of naloxone and opioid-induced side effects (nausea, vomiting, pruritus) were reduced by naloxone at both dose.

Naloxone and/or naltrexone at ultra-low doses may enhance the analgesic effects of opioids, enhance the antinociceptive effects of methadone, and decrease or block the development of opioid tolerance in rodents. The combination of oxycodone with an ultra-low dose of the antagonist naltrexone as a singular oral medication, Oxytrex, has been developed to prevent the development of tolerance in the treatment of moderate to severe chronic pain.

Aguado et. al. 2013 recently evaluated the effects of the opioid antagonist, naloxone, on remifentanil-induced tolerance or hyperalgesia in rats. Hyperalgesia was considered to be a decrease in mechanical nociceptive thresholds (von Frey), while opioid tolerance was considered to be a decrease in sevoflurane MAC reduction by remifentanil. An ultra-low dose of naloxone was able to block remifentanil-induced hyperalgesia and the MAC increase associated with hyperalgesia, but did not change opioid tolerance under inhaled anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who provide written informed consent.
* Age 18 years old or older (no upper age limit for inclusion)
* Gender: male or female.
* Surgery: Posterior spinal fusions

Exclusion Criteria:

* Allergy to opiates
* Chronic pain other than the primary indication for surgery
* Psychiatric illness
* History of substance abuse problem including alcohol &/or cannabis
* BMI > 35
* Subjects under 18 years of age.
* Subject without the capacity to give written informed consent. 8. Female subjects who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-02-25 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Occurrence of Opioid-induced hyperalgesia (OIH) | 24 hr Post-surgery
  Mechanical Pain Threshold-determined by von Frey filaments around the incision site
Occurrence of Opioid-induced hyperalgesia (OIH) | 48 hr Post-surgery
  Mechanical Pain Threshold-determined by von Frey filaments around the incision site

SECONDARY OUTCOMES:
Opioid consumption | 24 hr post surgery
  Opioid consumption required to control pain by Oral morphine equivalents
Opioid consumption | 48 hrs post surgery
  Opioid consumption required to control pain by Oral morphine equivalents
Cold Pressure Test | 24 hr post surgery
  Pain Threshold and Pain tolerance
Cold Pressure Test | 48 hrs post surgery
  Pain Threshold and Pain tolerance
Visual Analog Scale (VAS) Pain scores | Baseline
  VAS pain scores measured prior to surgery and at 4, 8 and 12h after extubation and again at 24h and 48h post-operatively
McGill short form questionnaire | Baseline
  The McGill questionnaire provides an assessment of pain quality and descriptors
Brief Pain Inventory | Baseline
  Brief Pain Inventory assesses both pain intensity and pain unpleasantness (the emotional component of pain is considered to be a better metric of subject satisfaction and quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Ariana Nelson, MD, Principal Investigator — Associate Clinical Professor
Locations (1):
- UC Irvine Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bekhit MH. Opioid-induced hyperalgesia and tolerance. Am J Ther. 2010 Sep-Oct;17(5):498-510. doi: 10.1097/MJT.0b013e3181ed83a0. PMID 20844348
- [Background] Lin SL, Tsai RY, Shen CH, Lin FH, Wang JJ, Hsin ST, Wong CS. Co-administration of ultra-low dose naloxone attenuates morphine tolerance in rats via attenuation of NMDA receptor neurotransmission and suppression of neuroinflammation in the spinal cords. Pharmacol Biochem Behav. 2010 Aug;96(2):236-45. doi: 10.1016/j.pbb.2010.05.012. Epub 2010 May 15. PMID 20478329
- [Background] King T, Ossipov MH, Vanderah TW, Porreca F, Lai J. Is paradoxical pain induced by sustained opioid exposure an underlying mechanism of opioid antinociceptive tolerance? Neurosignals. 2005;14(4):194-205. doi: 10.1159/000087658. PMID 16215302
- [Background] Vinik HR, Kissin I. Rapid development of tolerance to analgesia during remifentanil infusion in humans. Anesth Analg. 1998 Jun;86(6):1307-11. doi: 10.1097/00000539-199806000-00033. PMID 9620525
- [Background] Guignard B, Bossard AE, Coste C, Sessler DI, Lebrault C, Alfonsi P, Fletcher D, Chauvin M. Acute opioid tolerance: intraoperative remifentanil increases postoperative pain and morphine requirement. Anesthesiology. 2000 Aug;93(2):409-17. doi: 10.1097/00000542-200008000-00019. PMID 10910490
- [Background] Hansen EG, Duedahl TH, Romsing J, Hilsted KL, Dahl JB. Intra-operative remifentanil might influence pain levels in the immediate post-operative period after major abdominal surgery. Acta Anaesthesiol Scand. 2005 Nov;49(10):1464-70. doi: 10.1111/j.1399-6576.2005.00861.x. PMID 16223391
- [Background] Ma JF, Huang ZL, Li J, Hu SJ, Lian QQ. [Cohort study of remifentanil-induced hyperalgesia in postoperative patients]. Zhonghua Yi Xue Za Zhi. 2011 Apr 12;91(14):977-9. Chinese. PMID 21609550
- [Background] Cahill CM, Holdridge SV, Morinville A. Trafficking of delta-opioid receptors and other G-protein-coupled receptors: implications for pain and analgesia. Trends Pharmacol Sci. 2007 Jan;28(1):23-31. doi: 10.1016/j.tips.2006.11.003. Epub 2006 Dec 5. PMID 17150262
- [Background] Holdridge SV, Armstrong SA, Taylor AM, Cahill CM. Behavioural and morphological evidence for the involvement of glial cell activation in delta opioid receptor function: implications for the development of opioid tolerance. Mol Pain. 2007 Mar 12;3:7. doi: 10.1186/1744-8069-3-7. PMID 17352824
- [Background] Yalcin N, Uzun ST, Reisli R, Borazan H, Otelcioglu S. A comparison of ketamine and paracetamol for preventing remifentanil induced hyperalgesia in patients undergoing total abdominal hysterectomy. Int J Med Sci. 2012;9(5):327-33. doi: 10.7150/ijms.4222. Epub 2012 Jun 20. PMID 22745573
- [Background] Joly V, Richebe P, Guignard B, Fletcher D, Maurette P, Sessler DI, Chauvin M. Remifentanil-induced postoperative hyperalgesia and its prevention with small-dose ketamine. Anesthesiology. 2005 Jul;103(1):147-55. doi: 10.1097/00000542-200507000-00022. PMID 15983467
- [Background] Song JW, Lee YW, Yoon KB, Park SJ, Shim YH. Magnesium sulfate prevents remifentanil-induced postoperative hyperalgesia in patients undergoing thyroidectomy. Anesth Analg. 2011 Aug;113(2):390-7. doi: 10.1213/ANE.0b013e31821d72bc. Epub 2011 May 19. PMID 21596876
- [Background] Aguado D, Abreu M, Benito J, Garcia-Fernandez J, Gomez de Segura IA. Effects of naloxone on opioid-induced hyperalgesia and tolerance to remifentanil under sevoflurane anesthesia in rats. Anesthesiology. 2013 May;118(5):1160-9. doi: 10.1097/ALN.0b013e3182887526. PMID 23407105
- [Background] Kraemer WJ, Joseph MF, Volek JS, Hoffman JR, Ratamess NA, Newton RU, Fragala MS, French DN, Rubin MA, Scheett TP, McGuigan MR, Thomas GA, Gomez AL, Hakkinen K, Maresh CM. Endogenous opioid peptide responses to opioid and anti-inflammatory medications following eccentric exercise-induced muscle damage. Peptides. 2010 Jan;31(1):88-93. doi: 10.1016/j.peptides.2009.09.031. Epub 2009 Oct 2. PMID 19800931
- [Background] Luginbuhl M, Gerber A, Schnider TW, Petersen-Felix S, Arendt-Nielsen L, Curatolo M. Modulation of remifentanil-induced analgesia, hyperalgesia, and tolerance by small-dose ketamine in humans. Anesth Analg. 2003 Mar;96(3):726-732. doi: 10.1213/01.ANE.0000048086.58161.18. PMID 12598253
- [Background] Sen H, Sizlan A, Yanarates O, Emirkadi H, Ozkan S, Dagli G, Turan A. A comparison of gabapentin and ketamine in acute and chronic pain after hysterectomy. Anesth Analg. 2009 Nov;109(5):1645-50. doi: 10.1213/ANE.0b013e3181b65ea0. PMID 19843803
- [Background] Xuerong Y, Yuguang H, Xia J, Hailan W. Ketamine and lornoxicam for preventing a fentanyl-induced increase in postoperative morphine requirement. Anesth Analg. 2008 Dec;107(6):2032-7. doi: 10.1213/ane.0b013e3181888061. PMID 19020155
- [Background] Lopez-Alvarez S, Mayo-Moldes M, Zaballos M, Iglesias BG, Blanco-Davila R. Esmolol versus ketamine-remifentanil combination for early postoperative analgesia after laparoscopic cholecystectomy: a randomized controlled trial. Can J Anaesth. 2012 May;59(5):442-8. doi: 10.1007/s12630-012-9684-x. Epub 2012 Mar 2. PMID 22383085
- [Background] Koppert W, Sittl R, Scheuber K, Alsheimer M, Schmelz M, Schuttler J. Differential modulation of remifentanil-induced analgesia and postinfusion hyperalgesia by S-ketamine and clonidine in humans. Anesthesiology. 2003 Jul;99(1):152-9. doi: 10.1097/00000542-200307000-00025. PMID 12826855
- [Background] Engelhardt T, Zaarour C, Naser B, Pehora C, de Ruiter J, Howard A, Crawford MW. Intraoperative low-dose ketamine does not prevent a remifentanil-induced increase in morphine requirement after pediatric scoliosis surgery. Anesth Analg. 2008 Oct;107(4):1170-5. doi: 10.1213/ane.0b013e318183919e. PMID 18806023